CLINICAL TRIAL: NCT01308411
Title: Using Exhaled Nitric Oxide to Step Down Inhaled Corticosteroid Therapy in Asthma
Brief Title: Predicting Steroid Response Using Exhaled Nitric Oxide
Acronym: PCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 10010
Record Dates: First submitted 2010-05-28; First posted 2011-03-04 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: Asthma; Inhaled Corticosteroids; Exhaled Nitric oxide; Airways inflammation; Step down; Predicting response
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50% reduction in ICS dose (Experimental): All patients will reduce their inhaled corticosteroid dose by 50%
  Interventions: Other: 50% step down reduction in inhaled corticosteroid dose

INTERVENTIONS:
Other: 50% step down reduction in inhaled corticosteroid dose — All participants will have their inhaled corticosteroid dose reduced by 50%

SUMMARY:
Asthma affects 6% of the UK population and costs the NHS 1 billion pounds per year. £473 million alone is spent on inhaled steroid treatment which is designed to reduce inflammation in the breathing tubes.

Unfortunately knowing whether a patient is on just the right amount of steroid treatment is difficult, as asthma is a variable disease and the measures currently used to decide on increasing or decreasing steroid treatment bare little resemblance to the actual amount of inflammation present. Doctors may not reduce treatment as swiftly as necessary if a patient's asthma is well controlled because of concern over asthma attacks; this can result in potential over treatment with inhaled steroids. Although steroid treatment is safe, side effects can occur, and costs are large, so a strategy helping avoid over treatment would be beneficial both to patients and to the NHS.

As the investigators can more accurately measure airway inflammation present in the breathing tubes, using a chemical called nitric oxide present in a patient's breath, the investigators might be able to more accurately predict which patients could safely reduce their steroid treatment. Measuring nitric oxide is simple, and involves breathing into a special machine (similar to a roadside breathalyser). In this study the investigators will measure nitric oxide in patients with well controlled asthma, and reduce their asthma treatment by 50%. The investigators will then follow up the patients and remeasure their nitric oxide. At the end of the study the investigators will see if measurements of nitric oxide predicted which patients could safely step down their treatment. If successful this could help reduce the overall cost to the NHS of inhaled steroids and reduce steroid associated side effects.

DETAILED DESCRIPTION:
The principal objective is to establish whether a baseline measurement of airway inflammation, as measured in exhaled breath, or a variation in this measurement over time, can predict which patients can safely step down their asthma treatment without experiencing a loss of asthma control.

This study is designed to show whether a policy utilising measurements of exhaled nitric oxide (present in the breath) in guiding asthma treatment will be feasible, and is worth testing in a future prospective study.

The secondary objectives are to establish if this approach is feasible, safe and cost effective, when compared to current clinical guidelines.

Asthma is defined by the presence of symptoms associated with variable airflow obstruction, airway inflammation and airway hyperresponsiveness. Inhaled corticosteroids are one of the most commonly used treatments in asthma, currently £473 million per year is spent on these medications alone in the UK. Guidelines recommend that treatment decisions are based on assessment of symptoms and airflow obstruction. However, as there is no clear relationship between symptom control, airflow obstruction and airway inflammation, there is a risk that patients can be over treated. In the U.K. 80% of patients with asthma are managed in primary care; assessment of airway inflammation is not applicable in this setting, and management relies on the assessment of peak flow and symptoms.

Recently the concentration of nitric oxide present in exhaled breath (FENO) has been evaluated as a tool for assessing asthma. FENO is elevated in patients with asthma, is reduced by treatment with inhaled corticosteroids(8) and correlates with airway inflammation measured using bronchial biopsies and induced sputum. It is particularly applicable for monitoring asthma in primary care as the test is easy to perform, provides an immediate result, and inexpensive portable monitors are now available. FENO appears to be a very specific, but not sensitive, marker of airway inflammation and using a low level of FENO to predict lack of treatable airway inflammation may be successful. Evidence from a study in children suggests that this strategy may be successful. However, most studies using FENO to guide ICS dose have not adopted this approach and have instead been randomised controlled trials using a step up/ down protocol whereby a high FENO leads to a step up in ICS dose, and a low FENO leads to a step down in dose. They have attempted to both reduce asthma exacerbations despite also trying to reduce steroid dose. These studies have not met their primary endpoints and have been reviewed in a Cochrane report. In the study by Shaw et al. a similar amount of ICS was used over the duration of the study in both the group managed by FENO and the control group; there was however a difference at the end of the study, with the FENO group using significantly less ICS. In the study by Smith et al. the daily dose of ICS was significantly lower at all time points, however the study results are not applicable as patients did not receive long acting β2 agonists, and the ICS dose in the control group was artificially inflated. These trials lend weight to the idea that utilising a step down approach to FENO and ICS may be successful. Importantly there was no significant difference in asthma exacerbation rates between control or treatment group in either study, suggesting that an approach utilising by FENO is inherently safe. Other studies support this supposition; one study suggested a close correlation between loss of asthma control and ICS reduction, and another study demonstrated that within 2 weeks of a reduction in ICS, FENO rises back to baseline, however exact cut off values for a simple step down strategy have never been sought, despite evidence that this would constitute the best approach.

Most patients are at step 2-3 of the asthma guidelines, receiving ICS doses of between 200-800mcgs, and are managed in primary care; guidelines for a 50% reduction in ICS at 3 months are based on sparse evidence. If a low FENO can identify patients who can step down their ICS treatment without a risk of worsening asthma, a strategy using FENO is likely to be adopted into current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years of age)
* diagnosis of asthma
* step 2, 3 or 4 on the BTS asthma guidelines.
* Well controlled asthma and good lung function, as defined as a Juniper asthma control score of < 1.5.
* Not oral steroids in the last 3 months.

Exclusion Criteria:

* Incapable of giving informed consent.
* Poor treatment concordance.
* Pregnant women.
* Extensive co-morbidity.
* Previous admission to ITU with asthma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Whether a baseline measurement of airway inflammation, as measured in exhaled breath, or a variation in this measurement over time, can predict which patients can safely step down their asthma treatment without experiencing a loss of asthma control. | visit 4 and visit 5
  The main outcome is whether a low FENO value at baseline or visit four or visit five, or variability from baseline in FENO, predicts which participants can successfully step down ICS dose without provoking increasing asthma symptom

SECONDARY OUTCOMES:
The secondary objectives are to establish if this approach is feasible, safe and cost effective, when compared to current clinical guidelines. | visit 2 and visit 5
  The secondary outcome will be whether a rise in FENO from baseline predicted a clinically important drop in spirometry, methacholine PC20 or change in differential induced sputum cell counts

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Shaw, Dr, Principal Investigator — University of Nottingham
Locations (1):
- Leicester Glenfield Hospital, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Wilson E, McKeever T, Hargadon B, Hearson G, Anderson J, Hodgson D, Bailey H, Meakin G, Thomas M, Pavord ID, Harrison T, Shaw D. Exhaled nitric oxide and inhaled corticosteroid dose reduction in asthma: a cohort study. Eur Respir J. 2014 Dec;44(6):1705-7. doi: 10.1183/09031936.00093614. Epub 2014 Aug 19. No abstract available. PMID 25142486